CLINICAL TRIAL: NCT02909829
Title: An Open-label, Randomized, Three-way, Crossover Study to Assess the Safety and Efficacy of Closed-loop Delivery With and Without Meal Detection Module and Conventional Pump Therapy in Regulating Glucose Levels After a Missed Bolus in Adolescents With Type 1 Diabetes in Inpatient Settings
Brief Title: Safety and Efficacy of Artificial Pancreas With and Without a Meal Detection Module on Glycemic Control in Adolescents With Type 1 Diabetes After a Missed Bolus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Ahmad Haidar, Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Missed Bolus 9h
Record Dates: First submitted 2016-09-01; First posted 2016-09-21 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Artificial Pancreas; Closed-Loop Delivery; Insulin; Adolescent; Missed Bolus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Closed Loop Delivery (Experimental): Insulin will be delivered by subcutaneous insulin infusion pump. Infusion rates will be changed manually every 10 minutes based on the computer generated recommendation infusion rates, calculated from the glucose levels measured by a real time sensor. The computer generated recommendations are based on a predictive algorithm. Participants will eat breakfast and bolus, then eat lunch and not bolus.
  Interventions: Device: Closed Loop Delivery
- Closed Loop Delivery with Meal Detection Module (Experimental): Insulin will be delivered by subcutaneous insulin infusion pump. Infusion rates will be changed manually every 10 minutes based on the computer generated recommendation infusion rates, calculated from the glucose levels measured by a real time sensor. The computer generated recommendations are based on a predictive algorithm with an overlying meal detection module which detects missed meals and will increase insulin infusion rates based on a predictive meal detection algorithm. Participants will eat breakfast and bolus, then eat lunch and not bolus.
  Interventions: Device: Closed Loop Delivery with Meal Detection Module
- Conventional Pump Therapy (Active Comparator): Insulin will be delivered by subcutaneous insulin infusion pump with participants usual infusion rate. Participants will eat breakfast and bolus as per usual, then eat lunch and not bolus.
  Interventions: Device: Conventional Pump Therapy

INTERVENTIONS:
Device: Closed Loop Delivery — Insulin will be delivered by subcutaneous insulin infusion pump. Infusion rates will be changed manually every 10 minutes based on the computer generated recommendation infusion rates, calculated from the glucose levels measured by a real time sensor. The computer generated recommendations are based on a predictive algorithm.
  Arms: Closed Loop Delivery
Device: Closed Loop Delivery with Meal Detection Module — Closed Loop Delivery with Meal Detection Module Insulin will be delivered by subcutaneous insulin infusion pump. Infusion rates will be changed manually every 10 minutes based on the computer generated recommendation infusion rates, calculated from the glucose levels measured by a real time sensor. The computer generated recommendations are based on a predictive algorithm with an overlying meal detection module which detects missed meals and will increase insulin infusion rates based on a predictive meal detection algorithm
  Arms: Closed Loop Delivery with Meal Detection Module
Device: Conventional Pump Therapy — Insulin will be delivered by subcutaneous insulin infusion pump with participants usual infusion rate
  Arms: Conventional Pump Therapy

SUMMARY:
Despite current treatments for type 1 diabetes, maintaining blood glucose levels within a good range is a difficult task. A primary source for poor glucose control in adolescents is skipping insulin boluses at mealtimes. Advances in glucose sensors have motivated the research towards closed-loop delivery systems to automatically regulate glucose levels. Closed-loop delivery (artificial pancreas) is composed of an insulin pump, a continuous glucose sensor and a dosing algorithm that calculates the insulin dose to infuse based on sensor readings. The performance of a closed-loop delivery after a missed bolus may be improved if the computer program that calculates the insulin is enhanced with a meal detection module. The meal detection module will automatically detect the meal (which had no bolus delivered), and signal the delivery of more insulin.

The aim of this study is to assess the safety and efficacy of a closed-loop delivery with and without meal detection module compared to conventional pump therapy in regulating post-prandial glycemic levels after omission of a meal bolus.

The primary hypothesis is that closed-loop delivery with no meal detection module will reduce the mean increase in postprandial glucose levels after a missed bolus compared to conventional pump therapy.

DETAILED DESCRIPTION:
Despite current treatments for type 1 diabetes, maintaining blood glucose levels within a good range is a difficult task. A primary source for poor glucose control in adolescents is skipping insulin boluses at mealtimes. Advances in glucose sensors have motivated the research towards closed-loop delivery systems to automatically regulate glucose levels. Closed-loop delivery (artificial pancreas) is composed of an insulin pump, a continuous glucose sensor and a dosing algorithm that calculates the insulin dose to infuse based on sensor readings. The performance of a closed-loop delivery after a missed bolus may be improved if the computer program that calculates the insulin is enhanced with a meal detection module. The meal detection module will automatically detect the meal (which had no bolus delivered), and signal the delivery of more insulin.

The aim of this study is to conduct a randomized, three-way, cross-over trial to compare the efficacy of closed-loop delivery, closed-loop delivery with a meal detection module, and conventional pump therapy. The study aims to compare these three interventions for 9 hours in adolescents with poorly controlled type 1 diabetes.

Each 9 hours will include two meals of different carbohydrate content, of which one will not have a carbohydrate-matched prandial bolus. This study will allow for the assessment of the safety and efficacy of closed-loop delivery with and without a meal detection module compared to conventional pump therapy in regulating post-prandial glycaemia.

The aim of this study is to assess the safety and efficacy of a closed-loop delivery with and without meal detection module compared to conventional pump therapy in regulating post-prandial glycemic levels after omission of a meal bolus.

The primary hypothesis is that closed-loop delivery with no meal detection module will reduce the mean increase in postprandial glucose levels after a missed bolus compared to conventional pump therapy.

The secondary hypotheses are:

1. Closed-loop delivery with meal detection module will reduce the mean increase in postprandial glucose levels after a missed bolus compared to conventional pump therapy.
2. Closed-loop delivery with meal detection module will reduce the mean increase in postprandial glucose levels after a missed bolus compared to closed-loop delivery with no meal detection module.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least 12 months. (The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.)
2. The participant will have been on insulin pump therapy for at least 3 months.
3. HbA1c 7.5% to 12%.
4. Self-reported or documented history of missed-bolus for meals during the previous 6 months.

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
2. Severe hypoglycemic episode within one month of screening.
3. Pregnancy.
4. Current use of oral glucocorticoid medication (except low stable dose). Stable doses of inhaled steroids are acceptable.
5. Known or suspected allergy to the trial products, including the meal content.
6. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
7. Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc.).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
AUCinc: The incremental area under the curve (as compared to pre-meal glucose value) of the postprandial glucose excursions for the lunch meal. | 0 - 240 min postprandial lunch meal

SECONDARY OUTCOMES:
AUCinc: The incremental area under the curve (as compared to pre-meal glucose value) of the postprandial glucose excursions: a. >10.0 mmol/L; b. >13.9 mmol/L; c. >16.7 mmol/L | 0 - 240 min postprandial lunch meal
Percentage of postprandial time of sensor glucose measurements spent: a. <3.9 mmol/L; b. between 3.9 and 7.8 mmol/L; c. between 3.9 and 10.0 mmol/L; d. >10.0 mmol/L; e. >13.9 mmol/L; f. >16.7 mmol/L. | 0 - 240 min postprandial lunch meal
Mean sensor glucose concentration. | 9 hours
Total insulin delivery | 9 hours
Glucose concentration as measured by CGM at 2 hours (120 min) post-meal. | 120 min postprandial lunch meal
Incremental glucose concentration as measured by CGM at 2 hours (120 min) post-meal. | 120 min postprandial lunch meal
Incremental postprandial peak of glucose concentration as measured by CGM. | 0 - 240 min postprandial lunch meal
Number of hyperglycemic events > 18.0mmol/L. | 0 - 240 min postprandial lunch meal
1. Glucose concentration as measured by CGM at 5 hours (300 min) post-meal. Glucose concentration as measured by CGM at 5 hours (300 min) post-meal | 300 min postprandial lunch meal

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No